CLINICAL TRIAL: NCT05493774
Title: Preliminary Exploration of Applying Multi-person Simulation Training to Improve Nurse-led Burn and Scald Nursing Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chimei Medical Center (Other)
Responsible Party: Principal Investigator, Ying-Li Lee, Principal Investigator, Chimei Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 11105-012
Record Dates: First submitted 2022-08-01; First posted 2022-08-09 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Virtual Reality; High Fidelity Simulation Training
Keywords: Virtual Reality; High Fidelity Simulation Training; Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Virtual reality
  Interventions: Other: Multi-person virtual reality simulation scenario training
- Control group (Active Comparator): High Fidelity Simulation Training
  Interventions: Other: Multi-person high-fidelity simulation scenario training

INTERVENTIONS:
Other: Multi-person virtual reality simulation scenario training — Using multi-person virtual reality simulation scenario training to evaluate the learning effectiveness of nursing care for emergency burn and scald patients.
  Arms: Experimental group
Other: Multi-person high-fidelity simulation scenario training — Using multi-person high-fidelity simulation scenario training to evaluate the learning effectiveness of nursing care for emergency burn and scald patients.
  Arms: Control group

SUMMARY:
The purpose of this study was to compare the learning performance of trainees before and after learning burns and scald nursing care by applying the burns and scald virtual reality (VR) training module multi-person interactive training in different places and the traditional training model with a high-fidelity patient.

DETAILED DESCRIPTION:
The clinical instructors, standard practice nurses, training content, and assessment process were the same for the experimental and control groups, except for the training methods of the interventions. A pre-recorded instructional video on burn care was provided to each participant one week prior to the experiment for self-study. The experiment procedure includes research description, pre-test and pre-test questionnaire (about 10 minutes), VR hands-on teaching or environment familiarization phase (about 10 minutes), multi-person simulation training (about 15 minutes) and post-test debrief (about 5 minutes), post-test and questionnaire (about 10 minutes). After completing all experiments, the collected data will be analyzed by the researcher using SPSS version 22.0 for descriptive, t-test, and other statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

1. people who are above 20 years old, with a nurse practitioner certificate and an ACLS or AHA certificate within the validity period.
2. people who are interested in learning the role of a team leader in burn and scald care.
3. people who have never used an interactive virtual reality (VR) environment device.

Exclusion Criteria:

1. people who are prone to vertigo or poor balance and are prone to motion sickness.
2. people with a history of epilepsy.
3. eye surgery or injury within the past 6 months.
4. people with facial wounds that prevent them from wearing VR glasses.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Change in knowledge of burn and scald nursing care scale | Pre- and post-instructional design (immediately before conducting and after completing simulation scenario training)
  There were 10 items to evaluate the participants' knowledge of the burn and scald nursing care scale. Each item had four response options. The total score ranged from 0 to 10 and a higher score indicates a higher level of knowledge of burn and scalds nursing care.
Change in motivation and attitude toward learning and personal self-efficacy scale | Pre- and post-instructional design (before conducting and immediately after completing simulation scenario training)
  The motivation and attitude toward learning and personal self-efficacy scale included 21 items. Each item was scored on a five-point Likert-type scale ranging from 1 (strongly disagree) to 5 (strongly agree). The total score ranged from 21 to 105 and a higher score indicated a positive motivation and attitude toward learning and a higher level of personal self-efficacy in burn and scald nursing care.
Self-reported measure of satisfaction of learning | Post-instruction (immediately after completing simulation scenario training)
  The satisfaction of learning scale included 9 items. Each item was scored on a five-point Likert-type scale ranging from 1 (strongly disagree) to 5 (strongly agree). The total score ranged from 9 to 45 and a higher score indicated a higher level of satisfaction with the learning intervention in burns and scald nursing care.

CONTACTS AND LOCATIONS:
Locations (1):
- Chi Mei Medical Center, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No